CLINICAL TRIAL: NCT06412263
Title: Determinants of Post-operative Pain and Quality of Life Following Root Canal Treatment: A Prospective Clinical Study
Brief Title: Post-operative Pain and QoL After RCT
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 295316; Protocol number: AC21057 (Other: NHS Health Research Authority); REC Number: 21/YH/0180 (Other: NHS Lothian); Project no.: 2021/0159 (Other: Lothian R&D)
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-05

CONDITIONS: Post-operative Pain; Quality of Life
Keywords: Post-operative pain; Root canal treatment; Root canal retreatment; QoL; PoQoL
MeSH Terms: conditions — Pain, Postoperative | interventions — Retreatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- With post-operative pain (Assessed at 24 hours, 48 hours, 7 days): Root canal treatment or retreatment performed either in single-visit or multiple-visit. Post-operative pain will then be assessed after instrumentation and obturation (completion) for multiple-visit and after obturation only for the single-visit treatment.
  Interventions: Procedure: Routine root canal treatment/ retreatment
- Without post-operative pain (Assessed at 24 hours, 48 hours, 7 days): Root canal treatment or retreatment performed either in single-visit or multiple-visit. Post-operative pain will then be assessed after instrumentation and obturation (completion) for multiple-visit and after obturation only for the single-visit treatment.
  Interventions: Procedure: Routine root canal treatment/ retreatment
- Post-operative quality of life affected (Assessed at 24 hours, 48 hours, 7 days): Quality of life after root canal treatment both after instrumentation and after treatment completed will be assessed at 24H, 48H, 7 days. Factors that will be looked at are the chewing ability, speaking ability, sleeping whether painkillers are required to sleep, ability to carry out daily functions, difficulty in social relations and the overall quality of life.
  Interventions: Procedure: Routine root canal treatment/ retreatment
- Post-operative quality of life unaffected (Assessed at 24 hours, 48 hours, 7 days): Quality of life after root canal treatment both after instrumentation and after treatment completed will be assessed at 24H, 48H, 7 days. Factors that will be looked at are the chewing ability, speaking ability, sleeping whether painkillers are required to sleep, ability to carry out daily functions, difficulty in social relations and the overall quality of life.
  Interventions: Procedure: Routine root canal treatment/ retreatment

INTERVENTIONS:
Procedure: Routine root canal treatment/ retreatment — It is a routine clinical procedure involving root canal treatment/ retreatment and pain assessment after the treatment

SUMMARY:
This study is a prospective clinical study, which evaluates pain following the completion of non-surgical root canal treatment and re-treatment cases. Additionally, the effect of the post-operative pain on the quality of life (QoL) is also evaluated. The main objectives are: To evaluate the (i) incidence of post-operative pain after RCT at 24 hours, 48 hours and 7 days, (ii) factors affecting the incidence of post-operative pain and (iii) patients' post- operative quality of life (PoQoL) at 24 hours, 48 hours and 7 days.

Patients who are deemed suitable for this study, screened by clinicians on duty during Restorative New Patient Clinics, will be invited to participate in this study. They will be given the Patient Information Sheet (PIS) at the beginning of the session and will be given time to decide on whether to participate in the study or not. Patients who have consented to participate in the study will provide a written consent prior to the start of the study. Following this, the pre-operative pain assessment will be performed by their respective clinicians, based on the approved questionnaire.

Following the completion of the root canal treatment, for both post-instrumentation and post-obturation, the patients will be called by the principle investigator for the post-operative pain assessment at 24 hours, 48 hours and 7 days. The post-operative quality of life (QoL) will also be assessed via the phone call, at the same three time points. These assessments will be made based on an approved questionnaire.

DETAILED DESCRIPTION:
This study is a prospective clinical study, which evaluates pain following the completion of non-surgical root canal treatment and re-treatment cases. The study is planned to take place from October 2021 until April 2022. Patient cohort would be patients referred to the Edinburgh Dental Institute for root canal treatment. Root canal treatment and re-treatment cases will be performed by Postgraduate Trainees (Years 1,2 and 3) in Endodontology and Prosthodontics, core trainees, specialist registrars in the Restorative Departments and staff members of the Restorative Department, Edinburgh Dental Institute.

Patients who are deemed suitable for this study, screened by clinicians on duty during Restorative New Patient Clinics, will be invited to participate in this study. They will be given the Patient Information Sheet (PIS) at the beginning of the session and will be given time to decide on whether to participate in the study or not. If a suitable patient happens to not have the PIS and consent form during the 1st treatment visit, the patient will be provided with the PIS and consent form during the 1st treatment visit and will be given up to 24H to decide on participating in the study or not. The pre-operative assessment, which will include pain assessment will be conducted as per normal routine prior to the commencement of RCT. At 24H (+/- 2H) the Principal Investigator will call the patient to follow-up. If the patient has agreed to participate in the study, the 24H post-operative pain and quality of life assessment will be conducted at the same time. Once patients have agreed to participate, they will be required to provide written consent which will be attached together with the PIS. On the first treatment day, patients will be required to answer a pre-operative pain assessment Questionnaire, which will be answered in the presence of the clinician treating the patient, before the commencement of RCT. The pain questionnaire is the combination of Numeric Rating Scale (NRS) and Modified Verbal Rating Scale (MVRS) adapted from previous published studies, with the addition of question on the presence of pre-operative pain duration. The pre-operative questionnaire will incorporate questions on pain intensity, the need, name and dosage of painkillers used by the patient on that day, and the last dose taken (in hours) as well as the duration of pain felt, as the longer the duration of pre-operative pain felt has been associated with higher incidence of post-operative pain. Also, pre-operative pain felt within the last 24 hours prior to root canal treatment has been associated with higher probability of post-operative pain. Following the completion of treatment, patients will be provided with post-operative pain assessment questionnaire, for the evaluation of post-operative pain. A copy of the pain questionnaire will be given to the patients which will be used as a guide when the pain history is obtained. This will be carried out verbally via phone by the main investigator of the study. Patients will not be required to return the forms to the institute.

In addition to pain evaluation, this Pain Questionnaire also incorporates the intake of painkillers taken. In the event that painkillers are taken by patients for pain control, patients are required to record the pain intensity before the consumption of painkillers, apart from recording the dosage and frequency of painkillers taken. Patients will be advised on the standard painkiller regimen as a post-operative instruction after the completion of RCT. Painkiller consumption is also an indirect measure of post-operative pain intensity, hence, that is why this has been added to the Pain Assessment Questionnaire. Apart from the pain assessment, post-operative quality of life post-treatment will also be assessed, based on a questionnaire. Patients will be given the liberty to pull out from the study at any time, throughout the duration of the study. Similarly, the investigator will also be able to remove patients from the study, throughout the duration of the study, in the event that the teeth being root-treated were faced with complications that may alter the accuracy of the study. Withdrawal or removal will be recorded in the 'Withdrawal/ Removal Form'.

ELIGIBILITY:
Inclusion Criteria:

* All teeth requiring primary root canal treatment (only 1 tooth per patient)
* All teeth requiring root canal re-treatment (only 1 tooth per patient)
* Age 18-100 years old (completely formed root apex)
* Permanent teeth
* Periodontal pocket depth < 4mm and with mobility within normal limits
* The ability to give informed consent

Exclusion Criteria:

* Surgical root canal treatment
* Patients on long term analgesics and steroids
* Primary teeth
* Teeth with procedural errors either being referred for the management or created during the procedure
* Traumatized teeth
* Teeth with open apices
* Periodontally involved teeth
* Cases with hypochlorite accident
* Short or extruded root canal obturation
* Cases whereby canal patency was not achieved

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Those who have completed non-surgical nerve treatment (root canal treatment) and re-do nerve treatment (root canal re-treatment) cases.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Post-operative pain (both post-instrumentation and post-obturation) | 5 November 2021 until May 2023
  This study assesses pain after root canal treatment at 24 hours, 48 hours and 7 days for both single-visit and multiple-visit treatment, based on the following pain instruments: i) Numeric Rating Scaling, scores 0-10 with score 0 as no pain, scores 1-3 as mild pain, scores 4-6 as moderate pain and scores 7-10 as severe pain and ii) Modified Verbal Rating scale with scores 0-3, whereby score 0 as no pain, score 1 as mild pain and no analgesics required, score 2 moderate pain which can be controlled by analgesics and score 3 as severe pain that cannot be controlled by analgesics.
Post-operative quality of life | 5 November 2021 until May 2023
  It also looks at how the pain felt affects the patients' quality of life (QoL), which looked specifically at: i) difficulties in chewing, ii) difficulties in speaking, iii) difficulties in sleeping, iv) difficulties in performing daily functions, v) difficulties in performing social relations, vi) overall effects on the QoL at 24 hours 48 hours and 7 days, answered as yes or no.
Pre-operative factors affecting the incidence of post-operative pain following root canal treatment | 5 November 2021 until May 2023
  Factors affecting post-operative pain at 24 hours, 48 hours, 7 days.

SECONDARY OUTCOMES:
Duration of post-operative pain | 5 November 2021 until May 2023
  The duration of post-operative pain will be measured within the 7 days post-treatment
Severity of post-operative pain | 5 November 2021 until May 2023
  The severity of post-operative pain will be measured based on the numeric rating scale (NRS) and modified verbal rating scale (MVRS) based on the pain severity, whereby severe pain on the NRS ranges from 7-10 and a score 3 on the MVRS. Additionally, the need for painkillers and whether the painkillers are affective in managing the pain felt will also be an indirect measure of pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: Natrah A Fuad, BDS, Principal Investigator — Edinburgh Dental Institute
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mijiritsky E, Lerman Y, Mijiritsky O, Shely A, Meyerson J, Shacham M. Development and Validation of a Questionnaire Evaluating the Impact of Prosthetic Dental Treatments on Patients' Oral Health Quality of Life: A Prospective Pilot Study. Int J Environ Res Public Health. 2020 Jul 13;17(14):5037. doi: 10.3390/ijerph17145037. PMID 32668778
- [Background] Pasqualini D, Corbella S, Alovisi M, Taschieri S, Del Fabbro M, Migliaretti G, Carpegna GC, Scotti N, Berutti E. Postoperative quality of life following single-visit root canal treatment performed by rotary or reciprocating instrumentation: a randomized clinical trial. Int Endod J. 2016 Nov;49(11):1030-1039. doi: 10.1111/iej.12563. Epub 2015 Nov 5. PMID 26468626
- [Result] Arias A, de la Macorra JC, Hidalgo JJ, Azabal M. Predictive models of pain following root canal treatment: a prospective clinical study. Int Endod J. 2013 Aug;46(8):784-93. doi: 10.1111/iej.12059. Epub 2013 Feb 12. PMID 23402273
- [Derived] Fuad NA, Philpott RJ, Cresta M. Post-operative pain as a risk factor for reduced quality of life after root canal treatment: A prospective clinical study. Saudi Dent J. 2025 Jun 18;37(4-6):21. doi: 10.1007/s44445-025-00006-1. PMID 40528109

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT06412263/Prot_SAP_ICF_000.pdf